CLINICAL TRIAL: NCT06986824
Title: A Pilot Study To Assess The Effect Of Antepartum Perineal Massage Using A Pelvic Wand On Labor Agency And Pelvic Health
Brief Title: Perineal Massage Using A Pelvic Wand During Pregnancy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Ethan Litman, Clinical Fellow in Obstetrics, Gynecology and Reproductive Biology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025P000062
Record Dates: First submitted 2025-05-14; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Related; Pelvic Floor Disorders; Obstetric; Injury; Patient Empowerment
MeSH Terms: conditions — Pelvic Floor Disorders; Wounds and Injuries; Patient Participation

STUDY DESIGN:
Intervention Model Description: This is a randomized study with an intention-to-treat analysis with an intervention and control arm.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): The intervention arm will receive standard of care education about the benefits of perineal massage and receive instruction to perform the massage three times weekly. They will then watch a 2-minute video to demonstrate proper use and cleaning of the device to assist with antepartum perineal massage. Trained study personnel will also be available to answer questions on proper use, storage, and cleaning. Participants will be provided with the pelvic wand at enrollment and asked to use the device at least three times weekly for 10 minutes beginning at enrollment until their hospitalization for birth. This frequency and duration are what is recommended by pelvic floor physical therapists and is their standard of care.
  Interventions: Device: Pelvic wand
- Control (No Intervention): The control arm will receive standard of care verbal education about the benefits of self-directed (or partner) manual perineal massage in the antepartum period and during the birthing process. They will be given the device after birth before hospital discharge.

INTERVENTIONS:
Device: Pelvic wand — Use of a pelvic wand to perform perineal massage
  Arms: Intervention

SUMMARY:
There is limited research on the optimal strategy to reduce obstetric laceration, postpartum urinary retention, and postpartum pelvic pain. In systematic reviews, clinician-directed massage of the perineal muscles at the time of birth and patient directed massage of the perineal muscles in the third trimester to inconsistently reduce the incidence of severe obstetric laceration.1,2 However, there is significant heterogeneity of these studies is due in large part to the lack of a standardized protocols and unpredictability of clinician availability to perform perineal massage around the time of birth.

The purpose of this study is to understand how perineal massage with a pelvic wand in late pregnancy and during labor influences one's sense of self-control over the labor process and birth experience.

DETAILED DESCRIPTION:
Study Overview and Design This is a randomized controlled, single-center study to assess the effect of the Intimate RoseTM Pelvic Wand device (Figure 1) on the birth experience.

Methods Recruitment We will enroll eligible adult pregnant patients who plan to give birth at BIDMC.

Randomization After providing consent, we will randomize participants in a 1:1 ratio to the intervention or control arm.

Enrollment and Antepartum Period The intervention arm will receive standard of care education about the benefits of perineal massage and receive instruction to perform the massage three times weekly. They will then watch a 2-minute video to demonstrate proper use and cleaning of the device to assist with antepartum perineal massage. Trained study personnel will also be avilable to answer questions on proper use, storage, and cleaning. Participants will be provided with the pelvic wand at enrollment and asked to use the device at least three times weekly for 10 minutes begining at enrollment until their hospitilization for birth. This frequency and duration are what is recommended by pelvic floor physical therapists and is their standard of care.

The control arm will receive standard of care verbal education about the benefits of self-directed (or partner) manual perineal massage in the antepartum period and during the birthing process. They will be given the device after birth before hospital discharge.

Participants will be told to call their primary obstetric provider if they experience any symptoms when using the device or doing manual massage.

Device Use on Labor & Delivery The intervention arm will be asked to utilize the device every hour for at least 5 minutes. The participant will utilize the device until the second stage of labor (the onset of pushing), at which point the provider or bedside nurse can assist the participant in performing the perineal massage, which is the current standard of care on the BIDMC labor and delivery unit.

The control arm will perform perineal massage if they choose; there will be no research interaction with control arm participants on Labor and Delivery. We will give the device to the control arm participants after birth and before discharge in their postpartum room. As with the intervention group, they will be given the 2-minute video to demonstrate propoer use and cleaning, and they will be given an opportunity to ask questions.

Device Use During the Postpartum Period All participants will be asked to use the device at least three times weekly for 10 minutes after they receive clearance from their obstetric provider at their six-week postpartum visit. Study staff will call the participants to remind them on the instructions for use that were previously supplied. Participants will be asked to use the device until 12 weeks postpartum.

Participant Questionaries Participants will be asked to track their use of the device or manual massage and to complete the following questionnaires to assess their birth experience prior to hospital discharge and pelvic floor dysfunction and urinary dysfunction to be assessed at time of enrollment, 6 weeks postpartum, and 3 months postpartum.

* At enrollment and after consent: Pelvic Floor Distress Inventory 20 and Female Sexual Function Index
* During birth hospitalization: Labor Agentry Scale and Pelvic Floor Distress Inventory 20
* Six weeks postpartum: Pelvic Floor Distress Inventory 20
* 12 weeks postpartum: Labor Agentry Scale, Pelvic Floor Distress Inventory 20, Female Sexual Function Index

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Plan to give birth at BIDMC
* Age ≥18 years old
* English language preference
* 32-36 weeks 'gestation

Exclusion Criteria:

* Contraindication to vaginal birth, active genital herpes infection, fetal anomaly requiring cesarean birth).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean score difference between the two arms on the Labor Agentry Scale | During hospitalization (assessed up to 5 days)
  A clinically significant difference is defined as a mean score difference of 10 points

SECONDARY OUTCOMES:
The average number of completed massage sessions prior to hospitalization | 6-8 weeks prior to birth event
  The average number of completed massage sessions measured by analyzing diary responses between enrollment and admission to the hospital for birth
The average number of completed massage sessions during hospitalization | 24-48 hours
  The average number of completed massage sessions measured by analyzing diary responses during birth hospitalization.
The average number of completed massage sessions postpartum | 6 weeks post birth time point
  The average number of completed massage sessions measured by analyzing diary responses in the postpartum period
Number of patients with postpartum urinary symptoms | 12 weeks postpartum
  Number of patients with postpartum urinary symptoms based on survey responses.
Number of patients with pelvic floor dysfunction in the postpartum period | 6 weeks postpartum and 12 week postpartum
  Number of patients with pelvic floor dysfunction based on survey responses using the Pelvic Floor Distress Inventory 20 Questionnaire (PFDI-20) Female Sexual Function Index (FSFI)
obstetric lacerations at time of delivery | During hospitalization (assessed up to 5 days)
  The number of patients with obstetric lacerations at time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Little, MD, Principal Investigator — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data may be shared on a case by case basis

REFERENCES:
- [Background] Eason E, Labrecque M, Wells G, Feldman P. Preventing perineal trauma during childbirth: a systematic review. Obstet Gynecol. 2000 Mar;95(3):464-71. doi: 10.1016/s0029-7844(99)00560-8. PMID 10711565
- [Background] Aasheim V, Nilsen ABV, Reinar LM, Lukasse M. Perineal techniques during the second stage of labour for reducing perineal trauma. Cochrane Database Syst Rev. 2017 Jun 13;6(6):CD006672. doi: 10.1002/14651858.CD006672.pub3. PMID 28608597
- [Background] Hodnett ED, Simmons-Tropea DA. The Labour Agentry Scale: psychometric properties of an instrument measuring control during childbirth. Res Nurs Health. 1987 Oct;10(5):301-10. doi: 10.1002/nur.4770100503. PMID 3671777